CLINICAL TRIAL: NCT02658734
Title: A Multicenter, Open-Label, Single-Arm, Phase IV Study of Trastuzumab Emtansine in Indian Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Treatment With Trastuzumab and a Taxane
Brief Title: A Study of Trastuzumab Emtansine in Indian Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Unresectable Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Treatment With Trastuzumab and a Taxane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML29662
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: HER2 Positive Breast Cancer, Metastatic Breast Cancer, Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (1):
- Trastuzumab emtansine (Experimental)
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine — 3.6 mg/kg intravenously (IV) over 30-90 minutes on day 1 of 21 day cycle, repeated every 3 weeks

SUMMARY:
This is a Phase IV, single-arm, multicenter, open-label clinical trial designed to assess the safety of trastuzumab emtansine in Indian patients with HER2-positive unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (mBC) who have received prior treatment with trastuzumab and a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Prospectively confirmed HER2-positive (i.e., IHC 3+ or IHC 2+ and gene amplified by fluorescence in situ hybridization [FISH] positive) as assessed on primary tumor and/or metastatic site
* Documented progression of unresectable, locally advanced, or mBC, determined by the investigator
* Left ventricular ejection fraction (LVEF) >/= 50% by echocardiogram (ECHO)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A negative serum Beta-Human Chorionic Gonadotropin (Beta-HCG) test for women of childbearing potential (premenopausal or not meeting the definition of postmenopausal i.e. >/= 12 months of amenorrhea), and women who have not undergone surgical sterilization (i.e., absence of ovaries and/or uterus)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate non-hormonal methods of contraception, including at least one method with a failure rate of <1% per year, during the treatment period and for at least 7 months after the last dose of study drug
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 7 months plus 90 days (a spermatogenesis cycle) after the last dose of study drug. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 7 months after the last dose of study drug.

Exclusion Criteria:

* Prior treatment with trastuzumab emtansine
* Prior treatment with lapatinib or lapatinib with capecitabine or non-comparable biologic or biosimilar of trastuzumab
* Peripheral neuropathy of Grade >/= 3 per the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE [version 4.03])
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, synchronous or previously diagnosed HER2-positive breast cancer, or cancers with a similar curative outcome as those mentioned above
* History of receiving any anti-cancer drug/biologic or investigational treatment within 21 days prior to enrollment except hormone therapy, which can be given up to 7 days prior to enrollment; recovery of treatment-related toxicity consistent with other eligibility criteria
* History of exposure to cumulative doses of anthracyclines, as defined in the protocol
* History of radiation therapy within 14 days of enrollment
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as a history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 2 months (60 days) before enrollment
* CNS only disease
* History of a decrease in LVEF to < 40% or symptomatic congestive heart failure (CHF) with previous trastuzumab treatment
* History of symptomatic chronic heart failure (New York Heart Association [NYHA] Classes II-IV) or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction or unstable angina within 6 months of enrollment
* Current dyspnea at rest due to complications of advanced malignancy or requirement for continuous oxygen therapy
* Current severe, uncontrolled systemic disease
* Pregnancy or lactation
* Concurrent, serious, uncontrolled infections or current known infection with human immunodeficiency virus (HIV) or active hepatitis B and/or hepatitis C. For patients who are known carriers of hepatitis B virus (HBV), active hepatitis B infection must be ruled out, based on negative serologic testing and/or determination of HBV DNA viral load per local guidelines
* Presence of conditions that could affect gastrointestinal absorption: malabsorption syndrome, resection of the small bowel or stomach, and ulcerative colitis
* History of intolerance (such as Grade 3-4 infusion reaction) or known hypersensitivity to trastuzumab or murine proteins or any component of the product
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- India (13):
  - Apollo Hospitals International Limited, Gandhinagar, Gujarat
  - Manipal Hospital; Department of Oncology, Bangalore, Karnataka
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital; Medical Oncology, North WEST Delhi, National Capital Territory of Delhi
  - Christian Medical College & Hospital; Medicine, Vellore, Tamil Nadu
  - Healthcare Global Enterprises Limited, Bangalore
  - Artemis Health Institute, Gūrgaon
  - Fortis Memorial Research Institute; Department of Medical Oncology & Haematology, Gūrgaon
  - Sir Gangaram Hospital; Medical Oncology, New Delhi
  - Max Super Speciality Hospital, New Delhi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centres across India.
Groups:
- Trastuzumab Emtansine: 3.6 mg/kg of trastuzumab emtansine was administered to participants intravenously (IV) over 30-90 minutes on day 1 of 21 day cycle and was repeated every 3 weeks.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine
Started | 70
Completed | 13
Not Completed | 57
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal of Consent | 16
Not completed — Disease Progression | 28

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled in the study.
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 70
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Severity of Adverse Events
Description: Adverse events (AEs) grading was completed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Participants
  Grade 1 | 53
  Grade 2 | 40
  Grade 3 | 18
  Grade 4 | 2
  Grade 5 | 12

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the treatment. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study were also considered as adverse events.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 90.0

3. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: SAEs were defined as any AE that fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/ birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 40

4. Secondary Outcome: Severity of SAEs as Per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Severity refered to the intensity of an AE (e.g., rated as mild, moderate, or severe, or according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Participants
  Grade 1 | 1
  Grade 2 | 13
  Grade 3 | 10
  Grade 4 | 3
  Grade 5 | 6

5. Secondary Outcome: Percentage of Participants With Non-Serious Adverse Events of Special Interest
Description: Non-serious AEs of special interest included cases of severe drug-induced liver injury and suspected transmission of an infectious agent by the study drug.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 2.9

6. Secondary Outcome: Laboratory Results Abnormalities
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Number of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Number of Participants
  Basophils - High: number analyzed (Participants) | 4
  Basophils - High | 1
  Basophils/Leukocytes - Low: number analyzed (Participants) | 13
  Basophils/Leukocytes - Low | 13
  Basophils/Leukocytes - High: number analyzed (Participants) | 53
  Basophils/Leukocytes - High | 6
  Monocytes - High: number analyzed (Participants) | 4
  Monocytes - High | 2
  Hematocrit - Low | 57
  Hematocrit - High: number analyzed (Participants) | 30
  Hematocrit - High | 1
  Lymphocytes/Leukocytes - Low: number analyzed (Participants) | 66
  Lymphocytes/Leukocytes - Low | 38
  Lymphocytes/Leukocytes - High: number analyzed (Participants) | 66
  Lymphocytes/Leukocytes - High | 19
  Monocytes/Leukocytes - Low: number analyzed (Participants) | 61
  Monocytes/Leukocytes - Low | 8
  Monocytes/Leukocytes - High: number analyzed (Participants) | 65
  Monocytes/Leukocytes - High | 21
  Neutrophils/Leukocytes - Low: number analyzed (Participants) | 58
  Neutrophils/Leukocytes - Low | 14
  Neutrophils/Leukocytes - High: number analyzed (Participants) | 64
  Neutrophils/Leukocytes - High | 13
  Other Cells - High: number analyzed (Participants) | 4
  Other Cells - High | 3
  Other Cells/Leukocytes - High: number analyzed (Participants) | 59
  Other Cells/Leukocytes - High | 6
  Erythrocytes - Low | 41
  Erythrocytes - High | 15
  Eosinophils/Leukocytes - Low: number analyzed (Participants) | 66
  Eosinophils/Leukocytes - Low | 33
  Eosinophils/Leukocytes - High: number analyzed (Participants) | 56
  Eosinophils/Leukocytes - High | 13
  Bilirubin - Low: number analyzed (Participants) | 69
  Bilirubin - Low | 5
  Bilirubin - High | 22
  Bicarbonate - Low: number analyzed (Participants) | 58
  Bicarbonate - Low | 4
  Bicarbonate - High: number analyzed (Participants) | 61
  Bicarbonate - High | 11
  Direct Bilirubin - High: number analyzed (Participants) | 69
  Direct Bilirubin - High | 27
  Blood Urea Nitrogen - Low: number analyzed (Participants) | 64
  Blood Urea Nitrogen - Low | 21
  Blood Urea Nitrogen - High: number analyzed (Participants) | 58
  Blood Urea Nitrogen - High | 10
  Chloride - Low: number analyzed (Participants) | 61
  Chloride - Low | 20
  Chloride - High: number analyzed (Participants) | 64
  Chloride - High | 30
  Lactate Dehydrogenase - Low: number analyzed (Participants) | 69
  Lactate Dehydrogenase - Low | 8
  Lactate Dehydrogenase - High: number analyzed (Participants) | 55
  Lactate Dehydrogenase - High | 52
  Protein - Low: number analyzed (Participants) | 66
  Protein - Low | 10
  Protein - High | 30
  Urea - Low | 21
  Urea - High: number analyzed (Participants) | 66
  Urea - High | 10
  Partial Thromboplastin Time - Low | 22
  Partial Thromboplastin Time - High | 37

7. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of Study Medication
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 8.6

8. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Modification of Study Medication
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Participants
  Dose Reduced | 1
  Drug Interrupted | 11

9. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Interruption of Study Medication
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 15.7

10. Secondary Outcome: Exposure to Study Drug
Description: Exposure to study drug was the amount of study drug received over time (weeks).
Time Frame: From cycle 1 up to approximately 3 years
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Weeks | 39.60 (32.00)

11. Secondary Outcome: Percentage of Participants With Drug-Induced Liver Injury Meeting Hy's Law Criteria
Description: Hy's law criteria for potential drug-induced liver injury included elevated aminotransferase enzymes (ALT/AST) with concurrent elevated serum total bilirubin, gross jaundice, clinical disability and the need for hospital care.
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of Participants | 0

12. Secondary Outcome: Percentage of Participants With Congestive Heart Failure
Time Frame: From cycle 1 up to approximately 3 years
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percetnage of Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percetnage of Participants | 0

13. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) as Measured by Echocardiogram
Time Frame: From baseline to every three cycles of treatment up to Cycle 39 Day 1, and at the 2-days post-treatment, safety follow-up visits 1 and 3
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Percentage of LVEF
  Baseline | 59.49 (3.33)
  Cycle 03 Day 1: number analyzed (Participants) | 62
  Cycle 03 Day 1 | 0.08 (3.26)
  Cycle 06 Day 1: number analyzed (Participants) | 51
  Cycle 06 Day 1 | 0.20 (4.50)
  Cycle 09 Day 1: number analyzed (Participants) | 39
  Cycle 09 Day 1 | 0.23 (3.76)
  Cycle 12 Day 1: number analyzed (Participants) | 34
  Cycle 12 Day 1 | 0.06 (4.24)
  Cycle 15 Day 1: number analyzed (Participants) | 24
  Cycle 15 Day 1 | 0.38 (4.40)
  Cycle 18 Day 1: number analyzed (Participants) | 20
  Cycle 18 Day 1 | 0.15 (5.98)
  Cycle 21 Day 1: number analyzed (Participants) | 14
  Cycle 21 Day 1 | 2.50 (3.78)
  Cycle 24 Day 1: number analyzed (Participants) | 13
  Cycle 24 Day 1 | 0.23 (2.89)
  Cycle 27 Day 1: number analyzed (Participants) | 10
  Cycle 27 Day 1 | -0.60 (3.86)
  Cycle 30 Day 1: number analyzed (Participants) | 6
  Cycle 30 Day 1 | -0.17 (1.33)
  Cycle 33 Day 1: number analyzed (Participants) | 5
  Cycle 33 Day 1 | -1.20 (2.39)
  Cycle 36 Day 1: number analyzed (Participants) | 1
  Cycle 36 Day 1 | 0 (NA) — The standard deviation couldn't be calculated from one participant
  Cycle 39 Day 1: number analyzed (Participants) | 1
  Cycle 39 Day 1 | 0 (NA) — The standard deviation couldn't be calculated from one participant
  Safety Follow-Up 1: number analyzed (Participants) | 18
  Safety Follow-Up 1 | 1.28 (3.80)
  Safety Follow-Up 3: number analyzed (Participants) | 16
  Safety Follow-Up 3 | 1.38 (4.00)

14. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was based on the best (confirmed) overall response (BOR). ORR was defined as the number (%) of participants with confirmed complete response (CR) or partial response (PR) where the confirmation was performed no less than 4 weeks after the criteria for response were first met.
Time Frame: From cycle 1 up to approximately 3 years
Population: ITT population included all participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Participants | 16

15. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of enrollment until the date of first documented progression of disease or the date of death (by any cause in the absence of progression) whichever occurred first.
Time Frame: From cycle 1 up to approximately 3 years
Population: ITT population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Months | 14.0 [8.0 to 17.0]

16. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of enrollment until the date of death due to any cause. Participants not known to have died at the time of final analysis were censored based on the last recorded date on which the subject was known to be alive.
Time Frame: From cycle 1 up to approximately 3 years
Population: ITT population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 70
Months | NA [25.00 to NA] — The median duration of OS was not estimable since the OS was not achieved.

ADVERSE EVENTS:
Time Frame: From cycle 1 up to approximately 3 years
Arm/Group | Trastuzumab Emtansine
All-Cause Mortality (participants affected / at risk) | 12/70
Serious Adverse Events (participants affected / at risk) | 28/70
Other Adverse Events (participants affected / at risk) | 51/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine (N=70)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 4 (4)
PYREXIA (General disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (2)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 2 (2)
HYDROCEPHALUS (Nervous system disorders) | 2 (2)
SEIZURE (Nervous system disorders) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine (N=70)
ANAEMIA (Blood and lymphatic system disorders) | 11 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 (11)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 5 (7)
VOMITING (Gastrointestinal disorders) | 4 (4)
ASTHENIA (General disorders) | 8 (9)
PAIN (General disorders) | 8 (8)
PYREXIA (General disorders) | 19 (28)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (8)
HAEMOGLOBIN DECREASED (Investigations) | 4 (9)
PLATELET COUNT DECREASED (Investigations) | 7 (9)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (8)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5)
DIZZINESS (Nervous system disorders) | 5 (7)
HEADACHE (Nervous system disorders) | 11 (13)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (9)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT02658734/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT02658734/SAP_001.pdf